CLINICAL TRIAL: NCT07249710
Title: Immediate Effects of Pain Neuroscience Education in Physiotherapy Students With Chronic Non-specific Low Back Pain: a Pre-Post Intervention Study
Brief Title: Pain Neuroscience Education in Physiotherapy Students With Chronic Non-Specific Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe ŞİMŞEK (Other)
Responsible Party: Sponsor-Investigator, Ayşe ŞİMŞEK, Research Assistant, PhD Student, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KBU-2025-2208
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Chronic Non-specific Low Back Pain; Physiotherapist Students
Keywords: low back pain; pain neuroscience education; physiotherapy; pain knowledge
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Neuroscience Education Group (Experimental): Single-group intervention arm receiving a 70-minute Pain Neuroscience Education session. Outcome measures were collected at baseline and immediately after the intervention.
  Interventions: Behavioral: Pain Neuroscience Education (PNE)

INTERVENTIONS:
Behavioral: Pain Neuroscience Education (PNE) — The program consists of a single 70-minute Pain Neuroscience Education (PNE) session, which includes explanations of pain neurophysiology, central sensitization, biopsychosocial pain concepts, and cognitive-behavioral factors influencing chronic pain. Delivered by a trained certified physiotherapist.

SUMMARY:
This study aims to examine the immediate effects of a single-session Pain Neuroscience Education (PNE) program in physiotherapy students who experience chronic non-specific low back pain. The PNE session focuses on explaining pain mechanisms, central sensitization, and the role of psychological, cognitive, and behavioral factors in chronic pain. Participants complete outcome measures assessing pain intensity, pain knowledge, pain catastrophizing, and kinesiophobia before and immediately after the intervention. The purpose of the study is to determine whether a brief educational session can produce immediate improvements in pain-related outcomes in a student population.

DETAILED DESCRIPTION:
This study is a retrospective registration of a completed pre-post interventional study conducted among undergraduate physiotherapy students with chronic non-specific low back pain. The objective of the research was to evaluate the immediate effects of a single-session Pain Neuroscience Education (PNE) program on pain intensity, pain knowledge, pain-related beliefs, pain catastrophizing, and kinesiophobia.

The PNE session lasted approximately 70 minutes and was delivered by a physiotherapist trained in pain neuroscience and the biopsychosocial model. The session covered pain neurophysiology, the distinction between acute and chronic pain, central sensitization, factors contributing to persistent pain, and the role of cognition, emotions, and behaviors in pain experiences.

Participants completed self-report outcome measures at two time points:

Baseline (pre-intervention)

Immediately after the intervention

Outcome measures included the Numeric Pain Rating Scale (NPRS), Revised Neurophysiology of Pain Questionnaire (RNPQ), Pain Catastrophizing Scale (PCS), and Tampa Scale for Kinesiophobia (TSK). The study followed a single-group design with no control group and no randomization.

The study was conducted between April and October 2025 at Karabük University, Turkey. Ethical approval was obtained from the Karabük University Non-Interventional Clinical Research Ethics Committee (Decision No: 2025/2208), and written informed consent was obtained from all participants prior to data collection.

The results of this research aim to contribute to the understanding of how pain neuroscience education may provide immediate benefits in young adults experiencing chronic non-specific low back pain, particularly within a physiotherapy student population. The findings may support the integration of pain education approaches in physiotherapy curricula and early clinical training programs.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate physiotherapy and rehabilitation students
* Chronic non-specific low back pain for at least 3 months
* Pain intensity ≥3/10 on the Numeric Pain Rating Scale in the last week
* willing to participate

Exclusion Criteria:

* History of back surgery within the last 6 months
* Presence of neurological, orthopedic, cardiac, or systemic chronic disease
* Current participation in any physiotherapy, exercise, or medical treatment for low back pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (Numeric Pain Rating Scale) | Baseline and immediately after the intervention
  Pain intensity was measured using the Numeric Pain Rating Scale (NPRS), a 0-10 scale where higher scores indicate greater pain. Participants report their average low back pain in the last week. In the NPRS, individuals were asked to verbally rate the severity of their pain on a scale from 0 to 10. The minimum clinically significant difference for the NPRS was reported as 2 points.
Pain Knowledge (Revised Neurophysiology of Pain Questionnaire - rNPQ) | Baseline and immediately after the intervention
  Pain knowledge was measured using the Revised Neurophysiology of Pain Questionnaire (rNPQ). Higher scores indicate deeper understanding of pain neurophysiology.
Pain Catastrophizing (Pain Catastrophizing Scale - PCS) | Baseline and immediately after the intervention
  Pain catastrophizing was measured using the Pain Catastrophizing Scale (PCS). The Likert-type scale consists of 13 items, with each item scored from 0 (strongly disagree) to 4 (strongly agree). The higher the total score, the higher the degree of negative and exaggerated thoughts about pain
Kinesiophobia (Tampa Scale of Kinesiophobia - TSK) | Baseline and immediately after the intervention
  Kinesiophobia was assessed using the Tampa Scale for Kinesiophobia (TSK). Higher scores reflect greater fear of movement and reinjury. The TSK has a total of 17 items, and each item is scored using a 5-point Likert scale ranging from 1 = "disagree" to 4 = "strongly agree." The total score ranges from 17 to 68, with higher scores indicating greater fear of injury.

CONTACTS AND LOCATIONS:
Overall Officials: AYŞE ŞİMŞEK, MSc, Study Director — Karabuk University
Locations (1):
- Karabük University Faculty of Health Sciences, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No